CLINICAL TRIAL: NCT07083310
Title: The Effect of Health Education Conducted Using Two Different Methods on Women's Knowledge of Breast Cancer, Health Beliefs, Mammography Self-Efficacy, and Participation in Screening Programs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Serpil Özdemir, Associate Professor, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00004646
Record Dates: First submitted 2025-07-01; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Breast - Female
Keywords: breast cancer; mammography; motivational interview
MeSH Terms: conditions — Breast Neoplasms | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Participants were randomized into two intervention groups and one control group using block randomization via a digital program (randomiser.org). Six letter combinations of "A," "B," and "C" were created and randomly assigned to 78 participants in blocks of 13. The sequence of combinations was predetermined (see Figure 3.5). Letters "A," "B," and "C" were assigned to the health education, control, and motivational interviewing groups, respectively.
Who Masked: Participant
Masking Description: "The study is single-blind; only the participants are unaware of their group assignment, while the investigators are informed."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Health Education Group (Experimental): Participants will receive structured education sessions focused on increasing knowledge about breast cancer, risk factors, and the importance of early screening.
  Interventions: Behavioral: Health Education
- Motivational Interviewing Group (Experimental): Participants will engage in one-on-one counseling sessions using motivational interviewing techniques to enhance motivation and reduce barriers to mammography screening.
  Interventions: Behavioral: Motivational Interviewing
- Control Group (No Intervention): Participants will not receive any intervention during the study period.

INTERVENTIONS:
Behavioral: Health Education — Structured group education focused on breast cancer awareness, risk reduction, and early detection.
  Other Names: Assign to Arm: Health Education Group
  Arms: Health Education Group
Behavioral: Motivational Interviewing — Individual counseling sessions using motivational interviewing to enhance screening behavior.
  Other Names: Motivational Interviewing group
  Arms: Motivational Interviewing Group

SUMMARY:
Breast cancer is the most common cancer among women worldwide and can be deadly if not found early. Screening tests like mammograms help find breast cancer early, which improves the chances of successful treatment. However, many women do not take part in regular screenings because of fear, lack of knowledge, or other barriers.

This study looks at two ways of teaching women about breast cancer and mammogram screening: traditional health education and a counseling approach called motivational interviewing. Motivational interviewing helps women feel more confident and motivated to get screened by talking about their concerns and encouraging positive decisions.

The goal is to see which method better increases women's knowledge about breast cancer, their beliefs about health, their confidence in getting mammograms, and their actual participation in screening programs. The results will help improve how we support women in taking care of their breast health.

DETAILED DESCRIPTION:
Breast cancer, detected in approximately 2.3 million people worldwide each year and resulting in 670,000 deaths, ranks first among cancers in women and accounts for 25% of all cancer cases in women. In Turkey, screening of 2.5 million women in 2025 revealed 36,000 new breast cancer diagnoses. Today, breast cancer is a priority and significant public health issue due to its high morbidity and mortality rates, along with associated economic impacts such as healthcare costs and workforce losses. Factors facilitating the widespread prevalence of breast cancer like an epidemic include rapid population aging, unhealthy lifestyle behaviors, insufficient or inaccessible screening programs, negative attitudes and beliefs leading to refusal of screening, delays in early diagnosis and treatment, lack of knowledge, and underutilization of primary and secondary prevention services. A projection estimates that by 2040, the number of breast cancer cases worldwide will reach nearly three million, with about one million deaths annually.

Early diagnosis of breast cancer is the most important factor in increasing survival rates. Delays in early diagnosis increase mortality and morbidity, reduce treatment success, and lower quality of life. The World Health Organization strongly recommends community-based screening programs including mammography for breast cancer control. Mammography is a proven, effective, and reliable method for early detection of breast cancer. Literature reports that increased participation in mammography screening significantly reduces advanced-stage breast cancer cases and mortality. Mammography screening is conducted free of charge every two years for women aged 40-69 within Turkey's National Breast Cancer Screening Program, as in many developed and developing countries worldwide.

The most effective strategy to combat breast cancer threatening women's health is to screen at least 70% of the at-risk female population every two years by mammography. Participation rates in mammography vary between 7% and 84% across different regions. In Northern Europe, Denmark, Finland, and the Netherlands report participation rates of 84.1%, 82.8%, and 80.8%, respectively. In Southern Europe, Italy reports 61.3%, Latin America's Brazil between 12-31%, and Malaysia in Asia between 7-25%. In Turkey, despite free mammography services, participation ranges between 41-55%, which is below the desired level. Therefore, especially in developing and less developed countries, implementing evidence-based, supportive, and encouraging interventions accepted by the general population is recommended to increase mammography participation.

Meeting women's information needs regarding breast cancer and screening, positively influencing health beliefs, attitudes, and behaviors, and improving mammography self-efficacy are key factors in increasing participation. Factors negatively impacting participation include limited access to screening, fear of examination, low risk perception, lack of knowledge, and negative attitudes and beliefs about screening. Even though women may be aware of early breast cancer detection, low education levels, poor self-efficacy, and lack of motivation contribute to low screening participation. The literature recommends various methods to motivate women and remove perceived barriers to mammography screening. In Turkey, face-to-face interventions, home visits, and various educational methods and tools have increased mammography participation to varying degrees. Studies show that face-to-face and online counseling about breast cancer and early detection raise women's knowledge and motivation, improve health beliefs and attitudes, increase perceived benefits and self-efficacy, decrease perceived barriers, and consequently increase mammography participation. However, despite various health education interventions improving knowledge, awareness, and positive attitudes, participation rates rarely exceed 70%. Thus, raising knowledge and awareness alone is insufficient, and increasing motivation for screening behavior is essential.

Motivational interviewing (MI) is often used to encourage desired health behaviors. MI is a client-centered approach that helps individuals recognize ambivalence, make informed decisions, and resolve issues by enhancing motivation for positive health behaviors. MI consists of four stages: engaging, focusing, evoking, and planning. These aim to stimulate motivation for change, strengthen belief in change, support sustainability, and develop concrete plans for behavior change. MI has been shown to increase mammography participation. For example, a nurse navigation program including MI significantly increased mammography participation among Syrian refugee women. A randomized controlled trial with 120 Iranian women reported that MI counseling positively affected breast cancer screening behaviors, though mammography participation increased only to 26%. Systematic reviews and meta-analyses indicate that MI interventions may increase participation in breast cancer screening programs. However, no study in Turkish populations has investigated the effect of MI on mammography participation. Furthermore, randomized controlled trials on MI and breast cancer screening participation remain limited in quantity and quality, highlighting the need for well-designed, adequately powered, standardized MI trials. Additionally, no study has compared traditional health education with MI-based education on participation rates in breast cancer screening programs.

Therefore, well-designed randomized controlled trials comparing traditional health education and MI-based health education on women's breast cancer knowledge, health beliefs, mammography self-efficacy, and screening participation are needed.

This study aims to evaluate the effects of health education and motivational interviewing-based health education on women's breast cancer knowledge, health beliefs, mammography self-efficacy, and participation in screening programs.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in the study

Being a woman aged between 40 and 69 years

Being literate

Registered at the Family Health Center where the study is conducted

Exclusion Criteria:

* Having a first-degree relative (mother/sister) with a history of breast cancer

Having had a mammogram in the last two years and/or regularly

Having been diagnosed with any type of cancer

Being pregnant

Being in the postpartum period

Having a physical communication impairment (e.g., hearing, speech)

Having a diagnosis of neuropsychiatric illness

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 78 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Mammography Screening Participation Rate | Within 6 months after education/motivational interviewing intervention
  The rate of participants who attend mammography screening within 6 months will be evaluated using health records and surveys.

SECONDARY OUTCOMES:
Breast Cancer Knowledge Level | Baseline and 1 month after intervention

IPD SHARING:
Plan to Share IPD: No